CLINICAL TRIAL: NCT01830075
Title: The Life InSight Application Study: the Role of an Assisted Structured Reflection on Life Events and Ultimate Life Goals to Improve Quality of Life of Cancer Patients
Brief Title: The Life InSight Application Study (LISA)
Acronym: LISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other); Janssen, LP (Industry)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: W12-143#12.17.0161
Record Dates: First submitted 2013-04-05; First posted 2013-04-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Quality of Life
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group receives care as usual.
- Consultations (Experimental): An intervention of two consultations with a spiritual counselor supported by an e-application.
  Interventions: Behavioral: Consultations

INTERVENTIONS:
Behavioral: Consultations — The patients receive two consultations with a spiritual counsellor. In these consultations life evens and life goals are discussed.
  Arms: Consultations

SUMMARY:
Background:

It is widely recognised that spiritual care plays an important role in physical and psychosocial well-being of cancer patients but there is little evidence based research on the effects of spiritual care. The investigators will conduct the first randomized controlled trial on spiritual care using a brief structured interview scheme supported by an e-application. The aim is to examine whether an assisted reflection on life events and ultimate life goals can improve quality of life of cancer patients.

Design:

Based on the findings of the investigators previous research, the investigators have developed a brief interview model that allows spiritual counselors to explore, explicate and discuss life events and ultimate life goals with cancer patients. To support the interview, the investigators created an e-application for a PC or a tablet. To examine whether this assisted reflection improves quality of life the investigators will conduct a randomized trial. Patients with advanced cancer not amenable to curative treatment options will be randomized to either the intervention or the control group. The intervention group will have two consultations with a spiritual counselor using the interview scheme supported by the e-application. The control group will receive care as usual. At baseline and one and three months after randomization all patients fill out questionnaires regarding quality of life, spiritual wellbeing, empowerment, satisfaction with life, anxiety and depression and health care consumption.

Discussion:

Having insight into one's ultimate life goals may help to cope with a life event such as cancer. This is the first randomized controlled trial to evaluate the role of an assisted structured reflection on ultimate life goals to improve patients' quality of life and spiritual well being. The intervention is brief and based on concepts and skills that spiritual counselors are familiar with, it can be easily implemented in routine patient care and incorporated in guidelines on spiritual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with advanced cancer not amenable to curative treatment.
* Life expectancy ≥ 6 months.

Exclusion Criteria:

* Karnofsky Performance Score < 60.
* Insufficient command of the Dutch language to fill out Dutch questionnaires.
* Current psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 months
  The EORTC QLQ C15 is a questionnaire developed to assess the quality of life of palliative cancer care patients.
Spiritual well being | 4 months
  FACIT-Sp-12: Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being; The 12-item Spiritual Well-Being Scale

SECONDARY OUTCOMES:
patients empowerment | 4 months
  Patient empowerment is becoming more and more important, both from health care professionals' and from patients' perspective. The patients in the intervention arm of our study will reconstruct a life story and also define their life goals and their intention for the future. This can lead to a feeling of more empowerment to undertake actions which are important to the patient. We will assess patients' empowerment with a Dutch version of the Pearlin Mastery Scale developed by Pearlin en Schooler (1978). The Pearlin Mastery Scale measures the extent to which individuals perceive themselves in control of forces that significantly impact their lives. It consists of a 7-item scale. In previous studies, the instrument yielded satisfactory psychometric properties.
spirituality | 4 months
  Furthermore, as time patients' view on spirituality can change over time due to the intervention, we will measure spirituality by the Spiritual Attitude en Interests List (SAIL), developed by the Helen Dowling Institute in the Netherlands. The SAIL is a multidimensional questionnaire for studying spiritual experiences of religious and nonreligious people. Mean Cronbach's alphas ranged in research from .73 to .86.

OTHER OUTCOMES:
anxiety and depression | 4 months
  Changes in patients' perspective on satisfaction with life will be measured by the Diener Satisfaction with Life Scale. Furthermore, asfeelings of anxiety and depression may come up when patients realize the limited amount of time that is left to achieve life goals, feelings of anxiety and depression will be measured by the Hospital Anxiety and Depression Scale.
patients' health consumption | 4 months
  Patients' health consumption is assessed according to a shortened and for this study adjusted version of the Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness.
patients'satisfaction with the intervention | 4 months
  Finally, we will explore patients' satisfaction with the intervention by a telephone interview using a study-specific topic list.
satisfaction with life | 4 months
  Changes in patients' perspective on satisfaction with life will be measured by the Diener Satisfaction with Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM Laarhoven, van, MD, PhD, Principal Investigator — Acadamic Medical Center
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Kruizinga R, Scherer-Rath M, Schilderman JB, Hartog ID, Van Der Loos JP, Kotze HP, Westermann AM, Klumpen HJ, Kortekaas F, Grootscholten C, Bossink F, Schrama J, Van De Vrande W, Schrama NA, Blokland W, De Vos FY, Kuin A, Meijer WG, Van Oijen MG, Sprangers MA, Van Laarhoven HW. An assisted structured reflection on life events and life goals in advanced cancer patients: Outcomes of a randomized controlled trial (Life InSight Application (LISA) study). Palliat Med. 2019 Feb;33(2):221-231. doi: 10.1177/0269216318816005. Epub 2018 Dec 5. PMID 30516096
- [Derived] Kruizinga R, Scherer-Rath M, Schilderman JB, Sprangers MA, Van Laarhoven HW. The life in sight application study (LISA): design of a randomized controlled trial to assess the role of an assisted structured reflection on life events and ultimate life goals to improve quality of life of cancer patients. BMC Cancer. 2013 Jul 26;13:360. doi: 10.1186/1471-2407-13-360. PMID 23889978